CLINICAL TRIAL: NCT02894008
Title: A Phase IIa Safety Study to Assess the Safety and Immunogenicity of a New Leishmania Vaccine Candidate ChAd63-KH
Brief Title: A Study of a New Leishmania Vaccine Candidate ChAd63-KH
Acronym: Leish2a
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of York (Other)
Collaborators: University of Khartoum (Other)
Responsible Party: Principal Investigator, Paul Kaye, Professor Paul Kaye, University of York
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-000369-22
Record Dates: First submitted 2016-08-01; First posted 2016-09-09 (Estimated); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Leishmaniasis, Cutaneous
MeSH Terms: conditions — Leishmaniasis, Cutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ChAd63- KH (Experimental): Single intramuscular dose of ChAd63-KH, 1 x10(10)vp or, following safety review, 7.5 x 10(10)vp in adults
  Interventions: Drug: ChAd63-KH
- ChAd63-KH (Experimental): Single intramuscular dose of ChAd63-KH, 1x10(10)vp or, following safety review, 7.5 x 10(10)vp in adolescents
  Interventions: Drug: ChAd63-KH

INTERVENTIONS:
Drug: ChAd63-KH — ChAd63-KH in adults and adolescents with persistent PKDL.

SUMMARY:
This is a study to assess the safety of a new candidate Leishmania vaccine ChAd63-KH in patients with persistent post kala azar dermal leishmaniasis (PKDL).

This is a Phase II trial in patients with PKDL, to assess the safety and compare the humoral and cellular immune responses generated by the candidate vaccine in patients, and observe any clinical changes in the disease over a 42 day period following vaccination.

Study design: Eight adult volunteers will receive 1x10(10)vp and the subsequent eight volunteers will receive 7.5 x10(10)vp. Adolescents will be vaccinated with either 1x10(10)vp or 7.5 x10(10)vp, to be determined by evaluation of all available data after DSMB & CTSC review.

DETAILED DESCRIPTION:
This is a study to assess the safety of a new candidate Leishmania vaccine ChAd63-KH in patients with persistent post kala azar dermal leishmaniasis (PKDL). With 95% of cases occurring in India, Bangladesh, Nepal, the Sudan and Brazil, visceral leishmaniasis (VL) is a disease of the poor. With an estimated 40,000 or more deaths annually, mostly children and young adults, VL ranks second only to malaria amongst parasitic infections for mortality, and as measured by DALYs lost, it ranks in the top ten infectious diseases globally. No effective vaccine has yet been developed for VL / PKDL despite significant research efforts.

The investigators have recently completed a successful first-in-human clinical trial of a new therapeutic vaccine for VL / PKDL (ChAd63-KH). This trial demonstrated safety of ChAd63-KH in healthy UK adult volunteers and immunogenicity against the two Leishmania antigens on par with that seen to other vaccine candidate antigens in clinical development for other diseases (e.g. malaria, HCV, Ebola). Following external peer review of the data generated during LEISH1, the investigators have been awarded further Wellcome Trust funding to progress this vaccine into Phase II clinical trials in patients with PKDL.

Study design: The first eight adult volunteers will receive 1x10(10)vp and, following DSMB and CTSC review, the subsequent eights adult volunteers will receive 7.5 x10(10)vp. Doses will be administered at a single time point. Adolescents will be vaccinated with either 1x10(10)vp or 7.5 x10(10)vp, to be determined by evaluation of all available data after DSMB & CTSC review.

Objectives:

1. To assess the safety of a new candidate Leishmania vaccine ChAd63- KH in patients with persistent PKDL.

   Secondary objectives:
2. To compare the humoral and cellular immune responses generated by the candidate vaccine in patients with persistent PKDL.
3. To observe any clinical changes in the cutaneous PKDL disease over a 42 day period following vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Adults

The volunteer must be:

* Aged 18 to 50 years on the day of screening
* Females must be unmarried, single, or widowed
* Willing and able to give written informed consent

Adolescents

* Aged 12 to 17 years on the day of screening
* Female adolescents must be unmarried
* Written informed consent must be obtained from a parent

All Participants

* Uncomplicated PKDL of > 6 month's duration
* Available for the duration of the study
* In otherwise good health as determined by medical history, physical examination, results of screening tests and the clinical judgment of a medically qualified Clinical Investigator
* Negative for malaria on blood smear
* Judged, in the opinion of a medically qualified Clinical Investigator, to be able and likely to comply with all study requirements as set out in the protocol
* Willing to undergo screening for HIV, Hepatitis B and Hepatitis C
* For females only, willing to undergo urinary pregnancy tests on the day of screening, on the day of vaccination (prior to vaccination) and 7 and 42 days after vaccination.

Exclusion Criteria:

The volunteer may not enter the study if any of the following apply:

* Has mucosal or conjunctival PKDL
* Has had treatment for PKDL within 21 days
* Is negative for antibodies in the RK39 strip test
* Receipt of a live attenuated vaccine within 60 days or other vaccine within 14 days of screening
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine or a history of severe or multiple allergies to drugs or pharmaceutical agents
* Any history of severe local or general reaction to vaccination as defined as

  * Local: extensive, indurated redness and swelling involving most of the antero-lateral thigh or the major circumference of the arm, not resolving within 72 hours
  * General: fever ≥ 39.5°C within 48 hours, anaphylaxis, bronchospasm, laryngeal oedema, collapse, convulsions or encephalopathy within 48 hours
* Females - pregnancy, less than 12 weeks postpartum, lactating or willingness/intention to become pregnant during the study and for 3 months following vaccination.
* Seropositive for hepatitis B surface antigen (HBsAg) or Hepatitis C (antibodies to HCV)
* Any clinically significant abnormal finding on screening biochemistry or haematology blood tests or urinalysis
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months
* Tuberculosis, leprosy, or malnutrition
* Any other significant disease, disorder or finding, which, in the opinion of a medically qualified Clinical Investigator, may either put the volunteer at risk because of participation in the study, or may influence the result of the study, or the volunteer's ability to participate in the study
* Unlikely to comply with the study protocol

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Safety | 90 days
  Safety of a new candidate Leishmania vaccine in patients with persistent PKDL, assessed by the occurrence of biochemical, haematological and physiological responses which meet the criteria for adverse events/serious adverse events as described in the clinical trial protocol (v1.55)

SECONDARY OUTCOMES:
Cellular immune responses | 90 days
  To compare the humoral and cellular immune responses generated by the candidate vaccine in patients with persistent PKDL.
Clinical changes in cutaneous PKDL disease | 42 days following vaccination
  To observe any clinical changes in the cutaneous PKDL disease over a 42 day period according to a clinical grading score following vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Musa, MBBS, Principal Investigator — University of Khartoum
Locations (1):
- Centre for Tropical Medicine, Doka, Gedarif, Sudan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Younis BM, Osman M, Khalil EAG, Santoro F, Furini S, Wiggins R, Keding A, Carraro M, Musa AEA, Abdarahaman MAA, Mandefield L, Bland M, Aebischer T, Gabe R, Layton AM, Lacey CJN, Kaye PM, Musa AM. Safety and immunogenicity of ChAd63-KH vaccine in post-kala-azar dermal leishmaniasis patients in Sudan. Mol Ther. 2021 Jul 7;29(7):2366-2377. doi: 10.1016/j.ymthe.2021.03.020. Epub 2021 Mar 27. PMID 33781913